CLINICAL TRIAL: NCT01671059
Title: A Multi-Center, Non-Interventional Study to Evaluate Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab (ACROSS)
Brief Title: A Non-Interventional Study Evaluating Rheumatoid Arthritis Participants Treated With Tocilizumab (RoActemra/Actemra)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28314
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Participants with rheumatoid arthritis (RA) receiving tocilizumab either as combination therapy or monotherapy through routine clinical practice.

SUMMARY:
This non-interventional study evaluated the use and efficacy of tocilizumab (RoActemra/Actemra) in participants with moderate to severe rheumatoid arthritis. Eligible participants initiated on tocilizumab treatment according to the approved label were followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) American College of Rheumatology (ACR) criteria
* Participants in whom the treating physician made the decision to commence tocilizumab treatment (in accordance with the local label); this could include participants who had received tocilizumab treatment within 8 weeks prior to the enrollment visit

Exclusion Criteria:

* Participants who had received tocilizumab more than 8 weeks prior to the enrollment visit
* Participants who had previously received tocilizumab in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever was longer) before starting treatment with tocilizumab
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with rheumatoid arthritis initiated on treatment with tocilizumab (RoActemra/Actemra)
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Serbia (8):
  - Institut Za Reumatologiju; Reumatologiju, Belgrade
  - Military Medical Academy; Clinic of Rheumatology, Belgrade
  - Belgrade
  - Institute of Rheumatology and Cardiovascular Diseases; Rheumatology, Niška Banja
  - Niška Banja
  - Clinical Center Voivodina; Clinic for Immunology and Nephrology, Novi Sad
  - Special hospital for rheumatic diseases Novi Sad, Novi Sad
  - Novi Sad

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 80
Completed | 75
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Enrolled participants.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.98)
Gender [Count of Participants; unit: Participants]
  Female | 67
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab 6 Months After Treatment Initiation
Time Frame: 6 months
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants | 93.75

2. Secondary Outcome: Percentage of Participants With Dose Modifications
Time Frame: 6 months
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants with RA receiving tocilizumab either as combination therapy or monotherapy through routine clinical practice.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants | 11.2

3. Secondary Outcome: Percentage of Participants Receiving Tocilizumab After Failing Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 73
percentage of participants | 81.35

4. Secondary Outcome: Percentage of Participants Receiving Tocilizumab After Failing Other Biologic Agents
Time Frame: Baseline
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants | 18.8

5. Secondary Outcome: Reasons for Dose Modifications
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
participants
  Low level of neutrophils | 1
  Adverse event | 3
  Other reason | 1
  Missing data | 1
  Unknown reason | 3

6. Secondary Outcome: Percentage of Participants With Dose Interruptions
Time Frame: 6 months
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants | 3.75

7. Secondary Outcome: Percentage of Participants Discontinued From Tocilizumab for Safety Versus Efficacy
Time Frame: 6 months
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants
  Adverse Event | 3
  Lack of Efficacy | 1

8. Secondary Outcome: Percentage of Participants on Tocilizumab Monotherapy at Study Entry
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 73
percentage of participants | 13.6

9. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR; in millimeters per hour [mm/hour]) and global health assessment (participant-rated global assessment of disease activity using 10-mm visual analog assessment [VAS]); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 2.78 [0.51 to 5.25]
  Monotherapy | 2.45 [0.63 to 5.00]

10. Secondary Outcome: Percentage of Participants on Combination Therapy Achieving a Response by European League Against Rheumatism (EULAR) Category
Description: Percentage of participants achieving a response by EULAR category, including moderate, good, or no response. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline <-1.2 with a DAS28 score ≤3.2; Moderate response: change from baseline <-1.2 with DAS28 scores >3.2 to ≤ 5.1 or >5.1, or a change from baseline <-0.6 to ≥-1.2 with DAS28 scores ≤3.2 and >3.2 to ≤5.1; No response: change from baseline <-0.6 to ≥-1.2 with DAS28 score >5.1, or a change from baseline ≥-0.6 with DAS28 scores ≤3.2, >3.2 to ≤ 5.1, or >5.1.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
percentage of participants
  Good response | 62.3
  Moderate response | 32.1
  No response | 5.7

11. Secondary Outcome: Percentage of Participants on Monotherapy Achieving a Response by European League Against Rheumatism (EULAR) Category
Description: as for outcome 10
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
percentage of participants
  Good response | 71.4
  Moderate response | 28.6
  No response | 0.0

12. Secondary Outcome: Simplified Disease Activity Index (SDAI)
Description: Simplified Disease Activity Index (SDAI) is an index for measuring disease activity in RA and has a good correlation with the DAS28. The index is calculated using the following formula: SDAI: swollen joint count (SJC28) + tender joint count (TJC28) + physician global assessment (PGA) (10 cm visual analogue scale [VAS]) + PhGA (10 cm VAS + C-Reactive Protein (CRP) in milligrams/liter (mg/L). VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Scores range from 0 to 86, with higher scores also indicating increased disease activity.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 6.69 [0.03 to 27.20]
  Monotherapy | 4.5 [1.3 to 20.00]

13. Secondary Outcome: Clinical Disease Activity Index (CDAI) Score
Description: Clinical Disease Activity Index (CDAI) is an index for measuring disease activity in RA. The index was calculated using the following formula: CDAI = number of swollen joints using the 28-joint count (SJC28) + number of tender joints using the 28-joint count (TJC28) + patient global assessment of disease (PGA) based on 10 centimeter [cm] Visual Analog Scale [VAS] + physician global assessment of disease (PhGA) based on 10 cm VAS. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total CDAI scores range from 0 to 76, with higher scores indicating increased disease activity.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 7.05 [0.00 to 27.00]
  Monotherapy | 6 [1.00 to 20.00]

14. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) Response
Description: ACR response was calculated based on total joint count evaluation and other clinical and laboratory assessments. A positive ACR20 response required at least a 20% improvement (reduction) compared to baseline in swollen joint count (28 joints) and tender joint count (28 joints) and at least 3 of the following 5 assessments: patient's global assessment of pain, participant's global assessment of disease activity (PGH), physician's global assessment of disease activity (PhGH) (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale); participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity); acute phase reactant (CRP or ESR). A reduction in the level of and acute phase reactants was considered an improvement. ACR50 and ACR70 require a 50% and 70% improvement from baseline, respectively.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
percentage of participants
  ACR20 Response: Combination therapy | 87.8
  ACR20 Response: Monotherapy | 100
  ACR50 Response: Combination therapy | 46.3
  ACR50 Response: Monotherapy | 66.6
  ACR70 Response: Combination therapy | 41.4
  ACR70 Response: Monotherapy | 33.3

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESIs)
Description: An AESI includes serious/medically significant infections; opportunistic infections; cases of elevated alanine aminotransferase (ALT) and aspartate aminotransferase (AST), in combination with either elevated bilirubin or clinical jaundice; suspected transmission of an infectious agent by the study drug; myocardial infarction /acute coronary syndrome; gastrointestinal perforations; malignancies; anaphylaxis / hypersensitivity reactions (including injection site reactions); demyelinating disorders; stroke; serious/medically significant bleeding events; or serious/medically significant hepatic events.
Time Frame: 6 months
Population: Enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants
  AE | 25
  SAE | 13.75
  AESI | 1.25

16. Secondary Outcome: Patient Global Assessment of Disease Activity Score
Description: The Patient Global Assessment of disease activity provides an overall assessment of how RA affects the participant using a visual analogue score, where 0 indicates they are managing very well and 100 indicates they are managing very poorly. A decrease in the score indicates improvement.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 15 [0 to 80]
  Monotherapy | 14 [0 to 30]

17. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ is a participant self-reported questionnaire for assessing the extent of the participant's functional ability. It consists of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question has 4 response options, ranging from 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The HAQ scale is an average of all the scores and ranges from 0 to 3, where higher scores represent higher disease activity.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 0.43 [0 to 2.13]
  Monotherapy | 0.43 [0.1 to 2.37]

18. Secondary Outcome: Visual Analogue Scale (VAS) for Fatigue
Description: The VAS-fatigue provides an overall assessment of the level of fatigue that the participant is experiencing using a visual analogue score, where 0 indicates no fatigue, and 100 indicates extreme fatigue. A decrease in the score indicates improvement.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 15 [0 to 70]
  Monotherapy | 11 [0 to 30]

19. Secondary Outcome: Visual Analogue Scale (VAS) for Morning Stiffness
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was as limber as he/she would be during a day involving typical activities. Morning stiffness was assessed on a 100 mm VAS, where 0= none and 100= very severe.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 10 [0 to 100]
  Monotherapy | 12 [0 to 30]

20. Secondary Outcome: Visual Analogue Scale (VAS) for Pain
Description: The VAS-Pain provides an overall assessment of the severity of pain that the participant is experiencing using a visual analogue score, where 0 indicates no pain and 100 indicates unbearable pain. A decrease in the score indicates improvement.
Time Frame: 6 months
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
units on a scale
  Combination therapy | 20 [0 to 80]
  Monotherapy | 20 [0 to 30]

ADVERSE EVENTS:
Time Frame: 6 months
Description: An adverse event is any unfavorable or unintended sign or symptom associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 11/80
Other Adverse Events (participants affected / at risk) | 11/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=80)
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Medication error (Injury, poisoning and procedural complications) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Oral herpes (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=80)
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Transaminases increased (Investigations) | 1
Thrombocytopenia (Investigations) | 1
Blood cholesterol increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
Gamma-Glutamyltransferase increased (Investigations) | 1
Tonsillitis (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Lack of drug effect (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.